## Comparison of the Effectiveness of USG and Palpation Guidance Steroid Injection in Patients With Plantar Fasciitis

## NCT04709484 - 01.08.2021

## **Statistical Analysis**

Statistical analyses were done using SPSS version 20 statistical software (IBM Corp., Armonk, NY). Average, standard deviation and frequency were used as descriptive statistical methods. Shapiro-Wilk and Kolmogorov-Smirnov tests were used to evaluate the distribution of numerical data. Since the data were not suitable for normal distribution, Mann-Whitney U test was used to measure the difference between the groups and Willcoxon test was used to measure the temporal process. Bonferroni test was used to detect important differences. Pearson Chi Square test was used for the differences between discrete variables. The results were evaluated at a 95% confidence interval and p <0.05 significance level.